CLINICAL TRIAL: NCT00433290
Title: Protocol F1J-MC-HMFG Duloxetine 60 to 120 mg Versus Placebo in the Treatment of Patients With Osteoarthritis Knee Pain
Brief Title: Duloxetine vs. Placebo in the Treatment of Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11198; F1J-MC-HMFG
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Results first posted 2009-08-24 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Osteoarthritis Knee Pain
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Duloxetine
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — duloxetine 30 mg every day (QD), by mouth (PO) for 1 week, then duloxetine 60 mg QD, PO for 6 weeks, followed by duloxetine 60 mg QD, PO for 6 weeks for responders or duloxetine 120 mg QD, PO for 6 weeks for non-responders
  Other Names: LY248686; Cymbalta
  Arms: A
Drug: Placebo — placebo every day (QD), by mouth (PO) for 13 weeks
  Arms: B

SUMMARY:
The primary purpose of this study is to determine if duloxetine reduces pain severity in patients with osteoarthritis knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients with osteoarthritis knee pain.

Exclusion Criteria:

* Serious cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other medical or psychiatric condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the course of the study.
* Previous exposure to duloxetine.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edison, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow, Russia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg, Sweden

REFERENCES:
- [Derived] Yue L, Wang J, Enomoto H, Fujikoshi S, Alev L, Cheng YY, Skljarevski V. The Clinical Relevance of Pain Severity Changes: Is There Any Difference Between Asian and Caucasian Patients With Osteoarthritis Pain? Pain Pract. 2020 Feb;20(2):129-137. doi: 10.1111/papr.12835. Epub 2019 Nov 20. PMID 31505082
- [Derived] Williamson OD, Schroer M, Ruff DD, Ahl J, Margherita A, Sagman D, Wohlreich MM. Onset of response with duloxetine treatment in patients with osteoarthritis knee pain and chronic low back pain: a post hoc analysis of placebo-controlled trials. Clin Ther. 2014 Apr 1;36(4):544-51. doi: 10.1016/j.clinthera.2014.02.009. Epub 2014 Mar 17. PMID 24650448
- [Derived] Hochberg MC, Wohlreich M, Gaynor P, Hanna S, Risser R. Clinically relevant outcomes based on analysis of pooled data from 2 trials of duloxetine in patients with knee osteoarthritis. J Rheumatol. 2012 Feb;39(2):352-8. doi: 10.3899/jrheum.110307. Epub 2011 Dec 1. PMID 22133624
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 128 | 128
Completed | 93 | 111
Not Completed | 35 | 17
Not completed — Adverse Event | 24 | 7
Not completed — Lack of Efficacy | 1 | 5
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Protocol Violation | 3 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Entry Criteria Not Met | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 128 | 128 | 256
Age Continuous [Mean (Standard Deviation); unit: years] | 63.16 (8.75) | 61.90 (9.20) | 62.53 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 107 | 196
  Male | 39 | 21 | 60
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
  Greece | 16 | 16 | 32
  Russian Federation | 62 | 65 | 127
  Sweden | 14 | 14 | 28
  Canada | 25 | 23 | 48
Nonsteroidal Anti-Inflammatory Drug (NSAID) Use [Number; unit: participants]
  No | 81 | 75 | 156
  Yes | 47 | 53 | 100
Race/Ethnicity [Number; unit: participants]
  African | 0 | 3 | 3
  Caucasian | 126 | 124 | 250
  East Asian | 0 | 1 | 1
  Hispanic | 2 | 0 | 2
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meters squared] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/meters squared | 29.44 (4.66) | 29.65 (4.52) | 29.55 (4.58)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 81.05 (13.73) | 80.55 (12.24) | 80.80 (12.98)
Brief Pain Inventory Average Pain [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 6.07 (1.39) | 6.14 (1.27) | 6.11 (1.33)
Clinical Global Impressions of Severity Scale (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
  units on a scale | 3.34 (1.21) | 3.34 (1.33) | 3.34 (1.27)
Duration of Osteoarthritis Pain Since Onset [Mean (Standard Deviation); unit: years] | 8.14 (7.64) | 6.74 (6.58) | 7.44 (7.15)
Duration of Osteoarthritis Since Diagnosis [Mean (Standard Deviation); unit: years] | 6.16 (5.88) | 5.62 (6.20) | 5.89 (6.04)
Height [Mean (Standard Deviation); unit: centimeters] | 165.99 (8.69) | 165.02 (7.99) | 165.51 (8.34)
Weekly Mean of 24 Hour Average Pain Severity [Mean (Standard Deviation); unit: units on a scale] — This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represents the weekly mean of the scores of the average pain severity over the last 24 hours.
  units on a scale | 6.02 (1.18) | 6.07 (1.26) | 6.04 (1.22)

OUTCOME MEASURES:

1. Primary Outcome: Change in Brief Pain Inventory (BPI) 24-hour Average Rating
Description: A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Changes are timepoint minus baseline.
Time Frame: Baseline, Week 4, Week 7, Week 13
Population: All randomized participants. Intent-to-treat analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 128 | 128
units on a scale
  Week 4 Change from Baseline (n=121, n=127) | -1.80 (0.16) | -1.12 (0.15)
  Week 7 Change from Baseline (n=106, n=119) | -2.47 (0.18) | -1.41 (0.17)
  Week 13 Change from Baseline (n=100, n=116) | -2.72 (0.20) | -1.88 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Null hypothesis=the difference in the BPI average pain score between the duloxetine and placebo treatment goups at the last visit of the treatment phase is zero; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for Week 4 Change from Baseline. Treatment effects and interaction effects were evaluated based on two-sided significance level of 0.05. No adjustments for multiple comparisons were made; Repeated Measures Model: Change=Treatment,NSAID use, Pooled Investigator, Visit, Baseline, Treatment*Visit, Baseline*Visit
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for Week 7 Change from Baseline. Treatment effects and interaction effects were evaluated based on two-sided significance level of 0.05. No adjustments for multiple comparisons were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for Week 13 Change from Baseline. Treatment effects and interaction effects were evaluated based on two-sided significance level of 0.05. No adjustments for multiple comparisons were made; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Values at 13 Week Endpoint in Patient Global Impression of Improvement (PGI-I)
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: 13 Weeks
Population: All randomized participants with at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 123 | 127
units on a scale | 2.85 (1.24) | 3.09 (1.08)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.164, ANCOVA; Model: PGI-Improvement=Treatment, Pooled Investigator, baseline severity and NSAID used for main effect p-values

3. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Physical Function Subscale
Description: The WOMAC index (pain, stiffness, physical function subscales) will be completed by the patient. The physical function subscale has 17 questions on physical function difficulties with every day tasks. Each question is answered using a 5-point Likert scale (0 to 4). The physical function subscale has a range of scores of 0 (none) to 68 (extreme).
Time Frame: Baseline and 13 Weeks
Population: All randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 118 | 126
units on a scale
  Baseline | 35.05 (9.63) | 36.82 (8.15)
  Change from Baseline | -13.78 (10.78) | -10.75 (10.98)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.016, ANCOVA — P-value for Change from Baseline (change = endpoint - baseline); Model: Change=Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-value

4. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale
Description: The WOMAC index (pain, stiffness, physical function subscales) will be completed by the patient. The pain subscale has 5 questions on pain associated with every day tasks. Each question is answered using a 5-point Likert scale (0 to 4). The pain subscale has a range of scores of 0 (none) to 20 (extreme).
Time Frame: Baseline and 13 Weeks
Population: All randomized participants with baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 123 | 127
units on a scale
  Baseline | 10.24 (2.47) | 10.35 (2.66)
  Change from Baseline | -4.27 (3.30) | -3.49 (3.89)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.068, ANCOVA — P-value for Change from Baseline. Change = Week 13 value minus baseline value; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-value

5. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale
Description: The WOMAC index (pain, stiffness, physical function subscales) will be completed by the patient. The stiffness subscale has 2 questions on stiffness associated with time of day (morning versus later in the day). Each question is answered using a 5-point Likert scale (0 to 4). The pain subscale has a range of scores of 0 (none) to 8 (extreme).
Time Frame: Baseline and 13 Weeks
Population: All randomized participants with baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 123 | 127
units on a scale
  Baseline | 4.27 (1.36) | 4.50 (1.34)
  Change from Baseline | -1.63 (1.66) | -1.36 (1.71)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.064, ANCOVA — P-value for Change from Baseline. Change = Week 13 value minus baseline value; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-value

6. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Weekly Mean of the 24-Hour Average Pain and Worst Pain Scores
Description: This assesses the weekly mean of the average pain and worst pain experienced over the last 24-hours. This is an ordinal scale with scores for each subscale (average pain and worst pain) ranging from 0 (no pain) to 10 (worst possible pain). Change = endpoint minus baseline.
Time Frame: Baseline and 13 Weeks
Population: All randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 124 | 126
units on a scale
  Baseline Weekly 24-Hour Average Pain | 6.05 (1.16) | 6.08 (1.26)
  Change in Weekly 24-Hour Average Pain | -2.39 (1.90) | -1.78 (1.86)
  Baseline Weekly 24-Hour Worst Pain | 7.58 (1.26) | 7.53 (1.21)
  Change in Weekly 24-Hour Worst Pain | -2.57 (2.10) | -2.05 (1.90)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA — P-value for Change in Weekly 24-Hour Average Pain. Change = endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-value
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.047, ANCOVA — P-value for Change in Weekly 24-Hour Worst Pain. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-value

7. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Clinical Global Impression of Severity (CGI-S)
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
Time Frame: Baseline and 13 Weeks
Population: All randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 123 | 127
units on a scale | -0.63 (0.95) | -0.32 (1.32)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-value

8. Secondary Outcome: Number of Participants Who Responded to Treatment at 13 Week Endpoint
Description: Response to treatment was defined as a ≥ 30% reduction from baseline to endpoint in Brief Pain Inventory (BPI) average pain score. The BPI measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: 13 Weeks
Population: Number of randomized participants with non-missing response values.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 127
participants | 79 | 56
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

9. Secondary Outcome: Mean Change From Baseline to 13 Week Endpoint in Medical Outcomes Study Short Form-36 (SF-36) Medical Component Summary (MCS), Physical Component Summary (PCS), and Domain Scores
Description: MCS and PCS scores=0-100 (higher scores indicate better health status). Domain scores:general health=5-25, physical functioning=10-30, Role-physical=4-8, Role-emotional=3-6, social functioning=2-10, bodily pain=2-11, vitality=4-24, mental health=5-30.
Time Frame: Baseline and 13 Weeks
Population: Number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 128 | 128
units on a scale
  Mental Component Summary Baseline (n=119, n=121) | 55.86 (10.00) | 54.47 (10.16)
  Mental Component Summary Change from Baseline | 0.35 (8.11) | 1.10 (8.30)
  Physical Component Summary Baseline (n=119, n=121) | 30.59 (7.37) | 28.70 (6.87)
  Physical Component Summary Change from Baseline | 7.26 (8.55) | 4.76 (7.93)
  Bodily Pain Baseline (n=121, n=124) | 5.77 (1.25) | 5.58 (1.22)
  Bodily Pain Change from Baseline | 1.64 (1.70) | 1.12 (1.76)
  General Health Baseline (n=120, n=122) | 17.02 (4.38) | 16.61 (4.28)
  General Health Change from Baseline | 1.15 (2.96) | 0.64 (3.18)
  Mental Health Baseline (n=121, n=124) | 24.13 (4.06) | 23.67 (4.17)
  Mental Health Change from Baseline | 0.64 (3.31) | 0.56 (3.46)
  Physical Functioning Baseline (n=120, n=125) | 17.48 (3.90) | 16.38 (3.58)
  Physical Functioning Change from Baseline | 2.95 (4.17) | 2.16 (3.76)
  Role-Emotional Baseline (n=121, n=125) | 5.05 (1.19) | 4.76 (1.26)
  Role-Emotional Change from Baseline | 0.35 (1.22) | 0.40 (1.22)
  Role-Physical Baseline (n=121, n=125) | 5.31 (1.44) | 4.96 (1.33)
  Role-Physical Change from Baseline | 1.03 (1.80) | 0.70 (1.66)
  Social Functioning Baseline (n=121, n=125) | 8.18 (1.76) | 7.78 (1.69)
  Social Functioning Change from Baseline | 0.44 (1.63) | 0.44 (1.74)
  Vitality Baseline (n=121, n=124) | 16.10 (3.84) | 15.43 (3.69)
  Vitality Change from Baseline | 1.04 (3.46) | 0.81 (3.03)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.897, ANCOVA — P-value for Mental Component Summary Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Physical Component Summary Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value for Bodily Pain Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.051, ANCOVA — P-value for General Health Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.508, ANCOVA — P-value for Mental Health Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.019, ANCOVA — P-value for Physical Functioning Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.415, ANCOVA — P-value for Role-Emotional Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value for Role-Physical Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.342, ANCOVA — P-value for Social Functioning Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.135, ANCOVA — P-value for Vitality Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-values

10. Secondary Outcome: Change From Baseline to 13 Week Endpoint in EuroQoL Questionnaire - 5 Dimension (EQ-5D)
Description: The EQ-5D is an assessment of one's overall health. Consists of 5 items. Patients choose 1 of 3 options that best describe the status of each item. The EQ-5D US based index scores range from -0.11 to 1.0 where a score of 1.0 indicates perfect health. A positive change from baseline indicates health improvement.
Time Frame: Baseline and 13 Weeks
Population: Number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 124
units on a scale
  Baseline | 0.68 (0.16) | 0.66 (0.16)
  Change from Baseline | 0.09 (0.16) | 0.08 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.209, ANCOVA — P-value for EQ-5D Change from Baseline. Change = Endpoint minus baseline; Model: Change=Treament, Pooled Investigator, NSAID use and Baseline for main effect p-value

11. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Beck Depression Inventory - II (BDI-II)
Description: A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: Baseline and 13 Weeks
Population: All randomized participants. Intent-to-treat analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 122 | 127
units on a scale
  Baseline | 4.29 (6.27) | 5.35 (6.59)
  Change from Baseline | -0.82 (4.23) | -1.25 (3.90)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.871, ANCOVA — P-value for Change from Baseline. Change = Week 13 value minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-value

12. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A)
Description: A 14-item questionnaire with 2 subscales: anxiety (7 items) and depression (7 items). Each item is rated on a 4-point scale (0 to 3), giving maximum scores of 21 for anxiety subscale. Scores of 11 or more are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.'
Time Frame: Baseline and 13 Weeks
Population: Number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 122
units on a scale
  Baseline | 4.26 (3.32) | 4.16 (3.52)
  Change from Baseline | -1.11 (2.36) | -0.69 (2.44)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.138, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline; Model: Change = Treatment, Pooled Investigator, NSAID use and Baseline for main effects p-value

13. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory (BPI) Severity: Worst Pain Score
Description: A self-reported scale that measures the severity of pain based on the worst pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline and 13 Weeks
Population: Number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 127
units on a scale
  Baseline | 7.49 (1.51) | 7.50 (1.33)
  Change from Baseline | -2.74 (2.22) | -1.94 (2.29)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

14. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Severity: Least Pain Score
Description: A self-reported scale that measures the severity of pain based on the least pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline and 13 Weeks
Population: Number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 127
units on a scale
  Baseline | 4.70 (1.80) | 4.63 (1.86)
  Change from Baseline | -1.95 (2.27) | -1.24 (2.40)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

15. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Severity: Average Pain Score
Description: A self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline and 13 Weeks
Population: Number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 127
units on a scale
  Baseline | 6.09 (1.38) | 6.16 (1.26)
  Change from Baseline | -2.54 (1.99) | -1.78 (2.10)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Path analysis was used to test null hypothesis that change in BPI average pain severity depends on improvement of BDI or HADS-A, versus improvement in BPI average pain severity is due to a direct analgesic effect of treatment and not dependent on improvement in depression or anxiety symptoms. Model:Change in BPI average pain score=a0+a1*treatment group+a2*change in BDI total+a3*change in HADS-A+a4*BL of BPI average pain+a5*BL of BDI total+a6*BL of HADS-A; Test type: Superiority or Other; p = 0.002, Regression, Linear — P-value for direct analgesic effect. The null hypothesis was tested by testing a1=0 versus a1≠0

16. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Severity: Pain Right Now Score
Description: A self-reported scale that measures the severity of pain based on the pain right now. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline and 13 Weeks
Population: The number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 127
units on a scale
  Baseline | 5.45 (1.96) | 5.36 (1.91)
  Change from Baseline | -2.57 (2.29) | -1.80 (2.39)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value for Change from Baseline. Change=Endpoint minus baseline

17. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference: General Activity
Description: A self-reported scale that measures the interference of pain in the past 24 hours for general acitivity. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: The number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 126
units on a scale
  Baseline | 4.70 (2.28) | 5.17 (2.18)
  Change from Baseline | -2.26 (2.49) | -1.92 (2.34)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.050, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

18. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference: Mood
Description: A self-reported scale that measures the interference of pain in the past 24 hours on mood. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: The number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 126
units on a scale
  Baseline | 3.35 (2.53) | 3.60 (2.64)
  Change from Baseline | -1.59 (2.79) | -1.72 (2.58)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.913, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

19. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference: Walking Ability
Description: A self-reported scale that measures the interference of pain in the past 24 hours on walking ability. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: The number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 126
units on a scale
  Baseline | 5.41 (2.26) | 5.54 (2.20)
  Change from Baseline | -2.63 (2.58) | -2.07 (2.61)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.066, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

20. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference: Normal Work
Description: A self-reported scale that measures the interference of pain in the past 24 hours on normal work. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: The number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 126
units on a scale
  Baseline | 4.77 (2.39) | 4.88 (2.26)
  Change from Baseline | -2.43 (2.49) | -1.56 (2.53)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

21. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference: Relations With Other People
Description: A self-reported scale that measures the interference of pain in the past 24 hours on relations with other people. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: The number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 126
units on a scale
  Baseline | 2.36 (2.53) | 2.37 (2.35)
  Change from Baseline | -1.16 (2.62) | -0.89 (2.15)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.260, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

22. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference: Sleep
Description: A self-reported scale that measures the interference of pain in the past 24 hours on sleep. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: The number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 126
units on a scale
  Baseline | 3.66 (2.73) | 4.02 (2.73)
  Change from Baseline | -1.91 (2.74) | -1.91 (2.77)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.489, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

23. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference: Enjoyment of Life
Description: A self-reported scale that measures the interference of pain in the past 24 hours on enjoyment of life. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: The number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 126
units on a scale
  Baseline | 3.10 (2.78) | 3.29 (2.73)
  Change from Baseline | -1.53 (2.74) | -1.23 (2.73)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.131, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

24. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory Interference: Average Interference
Description: A self-reported scale that measures interference of pain on average of the 7 questions assessing the interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The average Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline and 13 Weeks
Population: The number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 121 | 126
units on a scale
  Baseline | 3.91 (1.98) | 4.13 (1.95)
  Change from Baseline | -1.93 (2.05) | -1.62 (1.99)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.082, ANCOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

25. Secondary Outcome: Adverse Events Reported as Reason for Discontinuation
Time Frame: over 13 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 128 | 128
participants
  Nausea | 5 | 0
  Insomnia | 1 | 2
  Arthralgia | 2 | 0
  Asthenia | 2 | 0
  Constipation | 1 | 1
  Abdominal pain upper | 0 | 1
  Abnormal dreams | 1 | 0
  Anxiety | 1 | 0
  Atrial fibrillation | 0 | 1
  Diarrhoea | 1 | 0
  Drug intolerance | 1 | 0
  Dyspepsia | 1 | 0
  Ejaculation disorder | 1 | 0
  Erectile dysfunction | 1 | 0
  Haemorrhoids | 1 | 0
  Hot flush | 1 | 0
  Lethargy | 0 | 1
  Memory impairment | 1 | 0
  Palpitations | 1 | 0
  Pyelonephritis acute | 0 | 1
  Sleep disorder | 1 | 0
  Supraventricular tachycardia | 1 | 0

26. Secondary Outcome: Statisically Significant Change From Baseline to 13 Week Endpoint in Laboratory Analytes
Time Frame: Baseline and 13 Weeks
Population: Number of participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: Units/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 128 | 128
Units/Liter
  Alkaline Phosphatase Baseline (n=120,n=126) | 77.33 (22.91) | 75.90 (22.30)
  Alkaline Phosphatase Change from Baseline | 2.38 (15.74) | -3.43 (14.56)
  Aspartate Amino Transaminase (AST) Baseline | 22.61 (7.89) | 24.23 (11.10)
  AST Change from Baseline (n=117,n=124) | 1.44 (8.32) | -1.37 (7.26)
  Gammaglutamyl Transpeptidase (GGT) Baseline | 25.56 (17.56) | 30.55 (30.72)
  GGT Change from Baseline (n=120,n=126) | 5.33 (20.40) | -2.10 (19.12)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for Alkaline Phosphatase Change from Baseline. Change = Endpoint minus baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.010, ANOVA — P-value for AST Change from Baseline. Change = Endpoint minus baseline
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.023, ANOVA — P-value for GGT Change from Baseline. Change = Endpoint minus baseline

27. Secondary Outcome: Statisically Significant Change From Baseline to 13 Week Endpoint in Chloride
Time Frame: Baseline and 13 Week Endpoint
Population: Number of randomized participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: millimole per Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 120 | 126
millimole per Liter
  Baseline | 104.38 (2.26) | 104.18 (2.43)
  Change from Baseline | -0.83 (2.62) | -0.08 (2.66)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.042, ANOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

28. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Vital Signs - Heart Rate
Time Frame: Baseline and 13 Weeks
Population: Number of participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 123 | 127
beats per minute
  Baseline | 68.74 (6.72) | 69.73 (7.76)
  Change from Baseline | 2.55 (7.22) | 0.06 (6.47)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.005, ANOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

29. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Vital Signs - Blood Pressure
Time Frame: Baseline and 13 Weeks
Population: Number of participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 123 | 127
mm Hg
  Systolic Blood Pressure (SBP) Baseline | 132.20 (13.75) | 131.42 (16.13)
  SBP Change from Baseline | -1.03 (11.45) | 0.89 (12.93)
  Diastolic Blood Pressure (DBP) Baseline | 79.73 (8.27) | 79.83 (9.26)
  DBP Change from Baseline | 0.09 (7.99) | 0.45 (7.95)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.285, ANOVA — P-value for SBP Change from Baseline. Change = Endpoint minus baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.668, ANOVA — P-value for DBP Change from Baseline. Change = Endpoint minus baseline

30. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Vital Signs - Weight
Time Frame: Baseline and 13 Weeks
Population: Number of participants with a baseline and at least one non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 123 | 127
kilograms
  Baseline | 81.01 (13.63) | 80.49 (12.27)
  Change from Baseline | -0.65 (2.01) | 0.47 (1.94)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for Change from Baseline. Change = Endpoint minus baseline

31. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory - Average Pain Score in Nonresponders
Description: A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  Non-Responders were defined as patients with a <30% reduction from baseline to visit 4 (7 weeks) in Brief Pain Inventory (BPI) average pain score.
Time Frame: Baseline and 13 Weeks
Population: Number of participants who did not respond to treatment after 6 weeks of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 33
units on a scale
  Baseline | 5.30 (1.61)
  Change from Baseline | -0.76 (2.03)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p = 0.040, t-test, 2 sided

32. Secondary Outcome: Number of Nonresponders at Week 7 Who Responded at Week 13 Endpoint
Description: Response was defined as a >=30% reduction from baseline to endpoint in Brief Pain Inventory average pain score. Nonresponders were defined as participants with a <30% reduction from baseline to Visit 4 (7 Weeks) in Brief Pain Inventory average pain score.
Time Frame: 13 Weeks
Population: Number of randomized participants who were non-responders at Visit 4 (7 weeks) and with non-missing response values.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 33
participants | 9

33. Secondary Outcome: Adverse Events Reported as Reason for Discontinuation in Nonresponders
Description: Nonresponders were defined as participants with a <30% reduction from baseline to Visit 7 (7 weeks) in Brief Pain Inventory average pain score.
Time Frame: over 13 Weeks
Population: Number of randomized participants who were nonresponders at Visit 4 (7 weeks).
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 33
participants
  Arthralgia | 1
  Constipation | 1
  Nausea | 1

ADVERSE EVENTS:
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 3 | 2
Other Adverse Events (participants affected / at risk) | 64 | 41
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Duloxetine | Placebo
Atrial fibrillation (Cardiac disorders) | 0/128 (0) | 1/128 (1)
Supraventricular tachycardia (Cardiac disorders) | 1/128 (1) | 0/128 (0)
Drug intolerance (General disorders) | 1/128 (1) | 0/128 (0)
Pyelonephritis acute (Infections and infestations) | 0/128 (0) | 1/128 (1)
Memory impairment (Nervous system disorders) | 1/128 (1) | 0/128 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Duloxetine | Placebo
Abdominal discomfort (Gastrointestinal disorders) | 2/128 (2) | 0/128 (0)
Abdominal pain upper (Gastrointestinal disorders) | 6/128 (6) | 1/128 (1)
Constipation (Gastrointestinal disorders) | 11/128 (14) | 2/128 (2)
Diarrhoea (Gastrointestinal disorders) | 6/128 (7) | 3/128 (3)
Dry mouth (Gastrointestinal disorders) | 6/128 (6) | 1/128 (1)
Dyspepsia (Gastrointestinal disorders) | 2/128 (3) | 1/128 (1)
Flatulence (Gastrointestinal disorders) | 3/128 (3) | 1/128 (1)
Nausea (Gastrointestinal disorders) | 13/128 (14) | 3/128 (3)
Asthenia (General disorders) | 4/128 (5) | 0/128 (0)
Fatigue (General disorders) | 3/128 (3) | 1/128 (1)
Pyrexia (General disorders) | 3/128 (3) | 1/128 (1)
Gastroenteritis (Infections and infestations) | 2/128 (2) | 0/128 (0)
Gastroenteritis viral (Infections and infestations) | 0/128 (0) | 2/128 (2)
Influenza (Infections and infestations) | 2/128 (2) | 2/128 (2)
Nasopharyngitis (Infections and infestations) | 3/128 (3) | 1/128 (1)
Urinary tract infection (Infections and infestations) | 0/128 (0) | 2/128 (2)
Blood potassium increased (Investigations) | 2/128 (2) | 2/128 (2)
Weight decreased (Investigations) | 2/128 (2) | 0/128 (0)
Anorexia (Metabolism and nutrition disorders) | 3/128 (3) | 0/128 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4/128 (4) | 4/128 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3/128 (3) | 2/128 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/128 (1) | 2/128 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2/128 (2) | 0/128 (0)
Dizziness (Nervous system disorders) | 7/128 (9) | 2/128 (2)
Dysgeusia (Nervous system disorders) | 4/128 (4) | 1/128 (1)
Headache (Nervous system disorders) | 4/128 (4) | 5/128 (6)
Somnolence (Nervous system disorders) | 5/128 (6) | 3/128 (3)
Tremor (Nervous system disorders) | 2/128 (2) | 0/128 (0)
Abnormal dreams (Psychiatric disorders) | 2/128 (2) | 0/128 (0)
Anxiety (Psychiatric disorders) | 2/128 (2) | 0/128 (0)
Insomnia (Psychiatric disorders) | 6/128 (7) | 3/128 (3)
Sleep disorder (Psychiatric disorders) | 2/128 (2) | 0/128 (0)
Dysuria (Renal and urinary disorders) | 2/128 (2) | 0/128 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 2/128 (2) | 0/128 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 3/128 (3) | 0/128 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2/128 (2) | 2/128 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7/128 (7) | 0/128 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0/128 (0) | 2/128 (2)
Hot flush (Vascular disorders) | 2/128 (2) | 0/128 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days